CLINICAL TRIAL: NCT02001142
Title: Effect of Exercise on Novel Insulin Signaling Events in Human Muscle
Brief Title: Effect of Exercise on Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ADA 7-13-TS-35
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Insulin Sensitivity; Exercise; Metabolism
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Other: Exercise
- Sedentary Control (No Intervention)

INTERVENTIONS:
Other: Exercise — single session of exercise
  Arms: Exercise

SUMMARY:
One of the main objectives of this study will be to assess potential differences in important risk factors associated with Metabolic Syndrome in overweight adults who do not participate in a regular exercise program compared with overweight individuals who do exercise regularly. In addition, we will determine the effects of a single, modest session of exercise on the body's ability to control blood sugar and regulate fat metabolism in obese sedentary adults vs. obese adults who live a physically active lifestyle. Our study focuses on identifying mechanisms responsible for improved insulin action related to regular exercise and to provide novel targets for preventing and treating type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index [BMI] = 30-45 kg/m2, fasting blood glucose concentration must be < or = to125 mg/dl, Hematocrit > or = to 34%, all women must be pre-menopausal

Exclusion Criteria:

* pregnancy or actively breastfeeding, weight instability (> or = to ± 5 lbs in the past month) evidence of cardiovascular or metabolic diseases, taking medications know to affect lipid and/or glucose metabolism.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09-17 (Actual); Study Completion 2016-09-17 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 2-3 hours
  A hyperinsulinemic-euglycemic clamp will be used to assess peripheral insulin sensitivity. Insulin sensitivity will be calculated from the clamp data as the rate of glucose infusion during the steady state period of the clamp - divided by the plasma insulin concentration at this time (units: mg/uU/ml/min)

SECONDARY OUTCOMES:
Resting Metabolic Rate | 20-30 min
Meal Tolerance Test | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Clincal Research Unit, Ann Arbor, Michigan, United States